CLINICAL TRIAL: NCT04375137
Title: Correlation Between Oxidative Stress Markers and COVID-19 Severity Index
Brief Title: Correlation Between Oxidative Stress Status and COVID-19 Severity
Status: Completed | Type: Observational
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, Principal Investigator, Shahid Beheshti University of Medical Sciences
Other Study IDs: SBMU.12543
Record Dates: First submitted 2020-05-03; First posted 2020-05-05 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe COVID: patients with positive PCR or compatible CT admitted in ICU or intubated
  Interventions: Diagnostic Test: Oxidative Stress ELISA Kit
- Non-severe COVID-19: patients with positive PCR or compatible CT admitted in ward without hypoxia
  Interventions: Diagnostic Test: Oxidative Stress ELISA Kit
- Healthy Controls: Healthy controls with negative IgM/IgG for COVID-19
  Interventions: Diagnostic Test: Oxidative Stress ELISA Kit

INTERVENTIONS:
Diagnostic Test: Oxidative Stress ELISA Kit — Checking oxidative stress markers and redox system status

SUMMARY:
During the new COVID-19 pandemic physicians all over the world have faced different challenges .Oxidative stress is a probable cause of multi organ failure in this setting which never has been evaluated in COVID-19 infection to the best of knowledge.Present study aimed to evaluate oxidative stress marker and redox system status in different COVID-19 patients regarding the severity of involvement.

DETAILED DESCRIPTION:
Oxidative stress is a probable cause of multi organ failure in this setting which never has been evaluated in COVID-19 infection to the best of knowledge.Present study aimed to evaluate oxidative stress marker and redox system status in different COVID-19 patients regarding the severity of involvement. Demographic and lab data of 60 COVID-19 confirmed positive cases gathered .These patients divided in to two arms: 1- severe COVID-19 which were intubated or admitted in intensive care unit due to severe hypoxia 2- non-severe COVID-19 patients which were not hypoxic and admitted in ward with no need to invasive oxygenation. All patients had positive RT-PCR positive nasopharyngeal swab results for COVID-19 or Lung CT scan compatible with COVID-19. Malondialdehyde(MDA) , Biopterin, Neopterin, SOD, Glutathione levels would be checked by ELISA tests and compared between these two groups and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* positive RT-PCR COVID-19
* compatible lung CT with COVID-19

Exclusion Criteria:

* not signing informed consent
* using antioxidants
* using statins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Severe COVID:Hypoxic intubated Non-severe COVID: non-hypoxic in ward Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
MDA concentration | 2 weeks
  MDA x 2 ULN in severe COVID

SECONDARY OUTCOMES:
Biopterin concentration | 2 weeks
  Difference between severe and controls
Neopterin rate of increase | 2 weeks
  Difference between severe and controls

CONTACTS AND LOCATIONS:
Overall Officials: Dalili, Principal Investigator — SBMU
Locations (1):
- Nooshin Dalili, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No